CLINICAL TRIAL: NCT04105647
Title: A Brief Messaging Lifestyle Modification Program for Patients With Non-small Cell Lung Cancer - A Pilot Study
Brief Title: Lifestyle Modification Program for Lung Cancer Patients - A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW19-597-2
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cancer, Lung
Keywords: Lifestyle modification; physical activity; messages
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The control group will receive a face-to-face group session and a package of instant messages related to healthy living information, but no information on lifestyle-integrated exercise and physical activity.
  The experimental group will receive a face-to-face group session and a package of information on lifestyle-integrated exercise and physical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will receive a face-to-face group session and a package of healthy lifestyle instant messages, including lifestyle-integrated exercise and physical activity.
  Interventions: Behavioral: Lifestyle-integrated exercise
- Control group (Placebo Comparator): The control group will receive a face-to-face group session and a package of healthy lifestyle instant messages, but not related to lifestyle-integrated exercise and physical activity.
  Interventions: Behavioral: Healthy living information

INTERVENTIONS:
Behavioral: Lifestyle-integrated exercise — The experimental group will receive a face-to-face group session and a package of instant messages related to lifestyle-integrated exercise and physical activity. The lifestyle-integrated exercise is modified from Zero-time exercise. It focuses on four exercise domains that patients with lung cancer could be done at home, including breathing, balance, aerobic, strength, stretching exercises
  Other Names: Experimental group
  Arms: Experimental group
Behavioral: Healthy living information — The control group will receive a face-to-face group session and a package healthy living instant messages, but not related to lifestyle-integrated exercise and physical activity.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Lung cancer is one of the most common cancer diseases, globally and locally. Several health benefits of increased physical activity (PA) have been reported for people with cancer. PA plays a critical role across the cancer trajectory, from prevention through to post-diagnosis and has been proposed as an alternative for improving physical and psychosocial health outcomes, reducing cancer recurrence, and cancer-specific and all-cause mortality.

Although there are a variety of exercise intervention programs for cancer patients, those programs were quite intensive, requiring individuals to commit extra time and effort. Feeling of overwhelmed appointments, lack of time, other barriers, including high cost and limited access to facilities are the most frequently reported barriers that prevent people from starting and maintaining exercise. Hence, the investigators propose to use a brief messaging lifestyle modification intervention program to incorporating simple and easy-to-do patient-centred home-based lifestyle-integrated exercise into daily activities of patients with lung cancer. The aims are to increase patients' physical activity and improve their fatigue, emotion and quality of life, compared to the control group.

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancer, globally and locally. Patients with lung cancer are in a uniquely challenging situation in their disease, comorbidities, and treatment that may lead to worsened symptoms and many negative health consequences, including fatigue, irritability, and impaired daytime functioning.

Physical activity (PA) is defined as 'any bodily movement produced by skeletal muscle that results in energy expenditure'. Several health benefits of increased PA have been reported for people with cancer. PA plays a critical role across the cancer trajectory, from prevention through to post-diagnosis and has been proposed as an alternative for improving physical and psychosocial health outcomes, reducing cancer recurrence, and cancer-specific and all-cause mortality. Although there are a variety of exercise intervention programs for cancer patients, those programs were quite intensive, requiring individuals to commit extra time and effort. Most clinicians underutilise exercise therapy, regardless of its low-cost way to improve symptoms and potential health outcomes. Feeling of overwhelmed appointments, lack of time, other barriers, including high cost and limited access to facilities are the most frequently reported barriers that prevent people from starting and maintaining exercise. Low motivation, fear to exercise, lack of knowledge about benefits are the most common barriers of engaging in physical activity for cancer patients.

Hence, the current proposal is to use a brief messaging lifestyle modification intervention program to incorporating simple and easy-to-do patient-centred home-based lifestyle-integrated exercise (light to moderate physical activity) into daily activities of patients with lung cancer.

The investigators hypothesised that patients in the experimental group would display significantly higher increases in physical activity and improvements in fatigue, emotion and quality of life, compared to the control group.

The objectives are to examine the short-term clinical effects on impacts on fatigue, emotion and quality of life in patients with lung cancer, and to evaluate the feasibility of a brief lifestyle-integrated exercise program to increase physical activity by a pilot study with objective fitness and subjective questionnaire assessment, and focus group interviews.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above;
* Diagnosis with non-small cell lung cancer
* General condition stable, either is undergoing or finished treatment
* Able to speak and read Chinese
* Able to complete the self-administered questionnaire
* Able to use instant messages such as WhatsApp or WeChat
* Mental, cognitive and physically fit determined by the clinicians/investigators
* Signed informed consent

Exclusion Criteria:

* Pre-operative lung cancer
* Skeletal fragility
* Serious active infection
* Inability to walk
* Previously untreated symptomatic brain metastases
* Severe respiratory insufficiency
* Uncontrolled pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue level at 6 weeks | Baseline and 6 weeks
  measured by Brief Fatigue Inventory

SECONDARY OUTCOMES:
Change in physical activity at 6 weeks | Baseline and 6 weeks
  measured by International Physical Assessment Questionnaire - Short version
Change in health-related quality of life at 6 weeks | Baseline and 6 weeks
  measured by European Organisation for Research and Treatment of Cancer and lung module questionnaire
Change in functional level at 6 weeks | Baseline and 6 weeks
  measured by Functional Assessment Cancer Therapy - Lung (FACT-L) questionnaire
Change in anxiety and depression symptoms at 6 weeks | Baseline and 6 weeks
  measured by Hospital Anxiety and Depression Scale. Each item is answered on a 4-point scale (0-3). The scores for the seven questions on depression are added together to obtain a score ranged from 0 to 21. The higher score the more depressed. The scores for the seven questions on anxiety are added together to obtain a score ranged from 0 to 21. The higher score the more anxiety.
Change in insomnia level at 6 weeks | Baseline and 6 weeks
  measured by Insomnia Severity Index
Change in sleep quality at 6 weeks | Baseline and 6 weeks
  measured by Pittsburgh Sleep Quality Index
Change in excessive daytime sleepiness at 6 weeks | Baseline and 6 weeks
  measured by Epworth Sleepiness Scale. It is a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, though not necessarily every day. The scores for the eight questions are added together to obtain a score ranged from 0 to 24. The higher score the more sleepiness.
Change in activity level at 6 weeks | Baseline and 6 weeks
  measured by fitbits
Change in hand grips strength at 6 weeks | Baseline and 6 weeks
  measured by a dynamometer
Change in lower limb strength at 6 weeks | Baseline and 6 weeks
  assessed by using a 30-second chair stand test to record the number of stands from chair in 30 seconds
Change in balance at 6 weeks | Baseline and 6 weeks
  assessed by a single-leg-stance test by recording the time within which the individual could effectively achieve balance on one leg
Change in flexibility at 6 weeks | Baseline and 6 weeks
  assessed by chair sit and reach test
Change in endurance at 6 weeks | Baseline and 6 weeks
  assessed by 6-minute walk

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Lai, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Agnes, Hong Kong
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The patient consent did not include sharing personal information to other researchers

REFERENCES:
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Peddle-McIntyre CJ, Singh F, Thomas R, Newton RU, Galvao DA, Cavalheri V. Exercise training for advanced lung cancer. Cochrane Database Syst Rev. 2019 Feb 11;2(2):CD012685. doi: 10.1002/14651858.CD012685.pub2. PMID 30741408
- See also: American Lung Association - Lung Cancer — https://www.lung.org/lung-health-and-diseases/lung-disease-lookup/lung-cancer/resource-library/lung-cancer-fact-sheet.html